CLINICAL TRIAL: NCT05732324
Title: Comparison of Percutaneous Coronary Intervention Optimization With Fractional Flow Reserve Versus Intravascular Ultrasound in the Treatment of Long Coronary Artery Lesions
Status: Completed | Type: Observational
Sponsor: Vilnius University Hospital Santaros Klinikos (Other)
Collaborators: Vilnius University (Other)
Responsible Party: Principal Investigator, Povilas Budrys, Principal Investigator, Vilnius University Hospital Santaros Klinikos
Other Study IDs: 19C1252
Record Dates: First submitted 2023-02-07; First posted 2023-02-17 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Coronary Artery Disease; Myocardial Ischemia; Myocardial Infarction
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Ischemia; Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- IVUS PCI optimization group: PCI will be optimized according to the IVUS. IVUS will be performed before PCI and will be used to select PCI strategy.
  Operators will try to reach an optimal anatomical PCI result as assessed by IVUS aiming for the following criteria:
  1. good stent apposition;
  2. good stent expansion (minimal stent area (MSA) >90% of distal reference lumen area and/or MSA ≥5.5mm2);
  3. plaque burden 5mm proximal and distal to the stent <50%);
  4. no stent edge dissection.
  After stent optimization an IVUS run will be performed. The IVUS run will be considered as final when further anatomical optimization will not be thought to be possible.
  Interventions: Procedure: IVUS guided PCI optimization; Diagnostic Test: FFR measurement
- Historical FFR PCI optimization group: The goal will be to achieve the optimal functional result, defined as an FFR post PCI ≥ 0.95. Further stented segment post-dilatation will be mandatory if FFR post PCI < 0.95. In case of a clear evidence of significant atheroma proximal or distal to the stented segment, the operators will be encouraged to optimize the functional result further by implanting additional stents.
  Interventions: Procedure: FFR guided PCI optimization; Diagnostic Test: FFR measurement

INTERVENTIONS:
Procedure: IVUS guided PCI optimization — PCI to long lesion will be optimized according to the IVUS.
  Groups: IVUS PCI optimization group
Procedure: FFR guided PCI optimization — PCI to long lesion will be optimized according to the FFR.
  Groups: Historical FFR PCI optimization group
Diagnostic Test: FFR measurement — Fractional flow reserve protocol will be applied for both FFR-guided and IVUS-guided PCI groups. FFR will be measured according to the standard practice using intravenous adenosine. FFR will be recorded before PCI at the distal third of the coronary artery and after PCI at the same location. In FFR optimization group more than one post PCI FFR measurements could be acquired if the operators performed additional optimization. In IVUS optimization group only one post PCI FFR measurement will be recorded after which the procedure will be considered to be finished, and no further interventions will be undertaken. The same FFR measurements will be performed at 9-12 months follow-up.

SUMMARY:
A single center, prospective, observational study to compare fractional flow reserve (FFR) and intravascular ultrasound (IVUS) percutaneous coronary intervention (PCI) optimization strategies on the functional PCI result (assessed with FFR) immediately post PCI and at 9-12 months after the treatment of long coronary artery lesions.

ELIGIBILITY:
Inclusion Criteria:

* Chronic coronary syndrome (stable angina; staged PCI to other lesions after acute myocardial infarction with ST segment elevation);
* Acute coronary syndrome without ST segment elevation (unstable angina or myocardial infarction without ST segment elevation);
* Functionally significant (FFR ≤ 0.8) lesion requiring a stent length of ≥ 30 mm and amenable for percutaneous coronary intervention.

Exclusion Criteria:

* Patient's age ≤ 18 years;
* Acute myocardial infarction with ST segment elevation;
* Treatment with dual antiplatelet therapy contraindicated;
* Survival expectancy ≤ 1 year;
* Known allergy to sirolimus, everolimus or zotarolimus.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with functionally significant long coronary artery lesions amenable to percutaenous coronary intervention.
Sampling Method: Probability Sample
Enrollment: 154 (Actual)
Dates: Start 2012-09-01 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
The rate of optimal functional PCI result | One year
  Post PCI FFR value < 0.9
The rate of poor functional PCI result | One year
  Post PCI FFR value ≤ 0.8
The rate of optimal anatomical PCI result | 1 day
  If all the four following IVUS criteria met: (1) good stent apposition; (2) good stent expansion (minimal stent area (MSA) >90% of distal reference lumen area and/or MSA ≥5.5mm2); (3) plaque burden 5mm proximal and distal to the stent <50%); (4) no stent edge dissection.

SECONDARY OUTCOMES:
The rate of target vessel failure (TVF) | One year
  Composite endpoint (target vessel related death (TV-death), target vessel related myocardial infarction (TV-MI), any target vessel revascularization (TV-R))

CONTACTS AND LOCATIONS:
Overall Officials: Giedrius Davidavicius, PhD, prof, Study Chair — Vilnius University Hospital Santaros Klinikos

IPD SHARING:
Plan to Share IPD: Undecided